CLINICAL TRIAL: NCT01064336
Title: Promacta Pregnancy Registry
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 113327; WE4032 (Other: GSK)
Record Dates: First submitted 2010-02-04; First posted 2010-02-08 (Estimated); Last update posted 2016-07-25 (Estimated); Status verified 2016-07

CONDITIONS: Purpura, Thrombocytopaenic, Idiopathic
Keywords: Thrombocytopenia; Pregnancy
MeSH Terms: conditions — Purpura; Thrombocytopenia | interventions — eltrombopag

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Pregnant women on eltrombopag: Any women with eltrombopag exposure during pregnancy that is reported prior to or after knowledge of the pregnancy outcome, substantiated by health care provider, and meeting the enrollment criteria: documentation that eltrombopag is being taken during pregnancy; timing of the prenatal exposure to eltrombopag (i.e. best estimation of which trimester in pregnancy that there was exposure to Eltrombopag for stratification and reporting purposes ); sufficient information to determine whether the pregnancy is being prospectively or retrospectively registered; whether the outcome of pregnancy was known at the time of the report; source of the report (i.e. health care professional, patient); full provider contact information to allow for follow-up (name, address, etc.)
  Interventions: Drug: Eltrombopag
- Infants: Infants through the first year of life whose mothers were exposed to eltrombopag during pregnancy.
  Interventions: Drug: Eltrombopag

INTERVENTIONS:
Drug: Eltrombopag — Eltrombopag is an orally bioavailable, small molecule thrombopoietin receptor (TPO-R) agonist for the treatment of idiopathic thrombocytopenic purpura

SUMMARY:
Since Idiopathic Thrombocytopenic Purpura (ITP) affects women who are of reproductive capacity and taking into account the lack of data concerning Eltrombopag (Promacta) use during pregnancy, the Eltrombopag (Promacta) Registry will be an essential component of the ongoing risk management for Eltrombopag (Promacta). The Registry will detect and record the events (live births, spontaneous abortions, stillbirths, elective terminations, therapeutic terminations, any serious pregnancy outcome, major and minor congenital anomalies, outcomes including preterm, small for gestation age, or intrauterine growth restriction adverse adverse effects on the following: immune system development, platelet number and function, neoplasm formation, bone marrow reticulin formation, thrombotic events) in the mother and/or the neonate/infant. The adverse events in the infant will be assessed through at least the first year of life. The Pregnancy Registry will compare the pregnancy and fetal outcomes of women exposed to eltrombopag Tablets during pregnancy to an unexposed control population. This study will be a prospective observational, exposure follow-up study.

DETAILED DESCRIPTION:
The outcomes of pregnancy are: live births, spontaneous abortions, stillbirths, elective terminations, therapeutic terminations, any serious pregnancy outcome, major and minor congenital anomalies, outcomes including preterm, small for gestation age, or intrauterine growth restriction adverse effects on the following: immune system development, platelet number and function, neoplasm formation, bone marrow reticulin formation, thrombotic events in the mother and/or the neonate/infant.

ELIGIBILITY:
Inclusion Criteria:

Documentation that Eltrombopag is being taken during pregnancy. Timing of the prenatal exposure to Eltrombopag (i.e. best estimation of which trimester in pregnancy that there was exposure to Eltrombopag for stratification and reporting purposes). Sufficient information to determine whether the pregnancy is being prospectively or retrospectively registered. Whether the outcome of pregnancy was known at the time of the report. Source of the report (i.e. health care professional, patient). Full provider contact information to allow for follow-up (name, address, etc.)

Exclusion Criteria: None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Women exposed to eltrombopag during pregnancy, as well as infants whose mothers were exposed to eltrombopag during pregnancy.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2010-03; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Outcome of Pregnancy (see Detailed Description for a complete list) | From exposure during pregnancy through at least the first year of infant's life

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline